CLINICAL TRIAL: NCT01038310
Title: Prognostic Value of FP-CIT-SPECT in Patients With Parkinson´s Disease
Brief Title: Prognostic Value of FP-CIT-SPECT in Parkinson´s Disease
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Joerg Spiegel, Assistant medical director, Universität des Saarlandes
Other Study IDs: JoergSpiegel2
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Parkinson´s Disease
Keywords: Parkinson´s disease; FP-CIT-SPECT
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators aim to study whether the nuclear medicine method FP-CIT-SPECT (more details see below) allows to predict the further clinical course of Parkinson´s disease. Especially the investigators are interested in the motor and cognitive functions of the parkinsonian patients.

DETAILED DESCRIPTION:
Background of this study:

Parkinson´s disease (PD) is a degenerative disorder of the nervous system. In PD, mainly the presynaptic dopaminergic neurons are affected: The dopamine synthesis as well as the active transport of dopamine into the synaptic gap by presynaptic dopamine transporters (DAT) is reduced. First parkinsonian symptoms occur when the concentration of dopamine within the basal ganglia is reduced by at least 80 per cent (Bernheimer et al. 1973). The reduced DAT density represents a typical phenomenon of PD. The DAT density can be measured by means of nuclear medicine methods: the tracer FP-CIT (Fluoropropyl-Carbomethoxy-Iodophenyl-Tropane) has a high affinity to presynaptic DAT (Booij et al. 1998). PD patients show a significantly lower striatal FP-CIT uptake than healthy controls. Therefore FP-CIT SPECT supports the diagnosis of PD (Benamer et al. 2000).

Aims of this study:

To test the predictive value of FP-CIT-SPECT concerning the clinical course of PD.

Study protocol:

In this study we now (time 2) examine 25 PD patients who where diagnosed as having PD and who underwent FP-CIT-SPECT in the years 2003 up to 2006 (time 1). At both times - time 1 and time 2 - the part III (motor part) of the Unified Parkinson´s Disease Rating Score (UPDRS-Score) was / will be performed in the "Off" state. Furthermore, at time 2 the CERAD examination will be performed. 25 patients have to be included, if a correlation coefficient r = 0.5, an error 1st order = 0.05 and an error 2nd order = 0.20 are assumed.

We intend to answer the following questions:

1. Is there a correlation between the DAT density - measured between 2003 and 2006 - and the then (time 1) clinical symptoms hypokinesia, rigidity, resting tremor, postural tremor (measured by the motor part of the UPDRS scale)?
2. Is there a correlation between the DAT density - measured between 2003 and 2006 - and the actual (year 2010, time 2) clinical symptoms hypokinesia, rigidity, resting tremor, postural tremor?
3. Is there a correlation between the DAT density - measured between 2003 and 2006 - and the change of clinical symptoms hypokinesia, rigidity, resting tremor, postural tremor 2003-2006 versus 2010 (delta = time 2 - time 1).
4. Is there a correlation between the DAT density - measured between 2003 and 2006 - and the actual (year 2010, time 2) cognitive functions (measured by the CERAD)?

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson´s disease according to the Queen Square Brain Bank criteria (Hughes et al. 1992).
* FP-CIT-SPECT at the Department of Nuclear Medicine, Saarland University, in the years between 2003 - 2006.
* Informed consent.

Exclusion Criteria:

* Severe neurological (except Parkinson´s disease), psychiatric or internal diseases after the FP-CIT-SPECT.
* Patients with a history of drug or alcohol abuse.
* Patients with dementia (Mini-Mental-State-Test < 24 points).
* Psychosis or antipsychotic treatment in the last 12 months.
* Patients with pallidotomy or deep brain stimulation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Parkinson´s disease who underwent FP-CIT-SPECT in the years between 2003 and 2006.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Correlation between striatal FP-CIT uptake (measured in the years 2003 - 2006) versus the then (time 1) and the actual (time 2) motor and cognitive functions. | Between 4 and 7 years after FP-CIT-SPECT

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Spiegel, Coordinator, Principal Investigator — Department of Neurology, Saarland University, Kirrberger Straße, D-66421 Homburg/Saar, Germany
Locations (1):
- Department of Neurology, Homburg/Saar, Saarland, Germany

REFERENCES:
- [Background] Bernheimer H, Birkmayer W, Hornykiewicz O, Jellinger K, Seitelberger F. Brain dopamine and the syndromes of Parkinson and Huntington. Clinical, morphological and neurochemical correlations. J Neurol Sci. 1973 Dec;20(4):415-55. doi: 10.1016/0022-510x(73)90175-5. No abstract available. PMID 4272516
- [Background] Booij J, Busemann Sokole E, Stabin MG, Janssen AG, de Bruin K, van Royen EA. Human biodistribution and dosimetry of [123I]FP-CIT: a potent radioligand for imaging of dopamine transporters. Eur J Nucl Med. 1998 Jan;25(1):24-30. PMID 9396871
- [Background] Benamer TS, Patterson J, Grosset DG, Booij J, de Bruin K, van Royen E, Speelman JD, Horstink MH, Sips HJ, Dierckx RA, Versijpt J, Decoo D, Van Der Linden C, Hadley DM, Doder M, Lees AJ, Costa DC, Gacinovic S, Oertel WH, Pogarell O, Hoeffken H, Joseph K, Tatsch K, Schwarz J, Ries V. Accurate differentiation of parkinsonism and essential tremor using visual assessment of [123I]-FP-CIT SPECT imaging: the [123I]-FP-CIT study group. Mov Disord. 2000 May;15(3):503-10. PMID 10830416
- [Background] Hughes AJ, Daniel SE, Kilford L, Lees AJ. Accuracy of clinical diagnosis of idiopathic Parkinson's disease: a clinico-pathological study of 100 cases. J Neurol Neurosurg Psychiatry. 1992 Mar;55(3):181-4. doi: 10.1136/jnnp.55.3.181. PMID 1564476